CLINICAL TRIAL: NCT04830293
Title: The Effect of Head Position During Thyroidectomy on Cerebral Oxygenation and Postoperative Cognitive Functions
Brief Title: Effect of Head Position During Thyroidectomy on Postoperative Cognitive Functions
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Aydin, associate professor doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2119-40-14/02
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Thyroid; Carotid Doppler; Cerebral Perfusion
Keywords: Head position; Cerebral Oxygenation; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Thyroid Diseases; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Carotis Doppler Ultrasound — Neck was rotated about 30-45 ° to the opposite side of the image. The common carotid artery and internal jugular vein were viewed transversely on the B Mode USG image. Then, the probe was rotated approximately 90 ° and the carotid artery was visualized in the longitudinal plane. The probe and guide line were adjusted so that the Doppler angle was 60 °. The image was created with the guiding line parallel to the blood flow. After imaging of the carotid artery bifurcation, measurements were made 1 cm distal to this level.

SUMMARY:
The aim of our study is to observe the effect of head-neck position of patients scheduled for thyroidectomy, on carotid artery blood flow, regional cerebral oxygen saturation measured using near-infrared spectroscopy technology, and postoperative cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* undergo a total thyroidectomy operation
* ASA I-II
* euthyroid patients in the preoperative period

Exclusion Criteria:

* Hemoglobin< 8 g / dl
* Hypertension
* Hyperlipidemia
* Pregnancy
* Patients diagnosed with diabetes mellitus
* Cerebrovascular insufficiency
* Known carotid artery lesion
* Metabolic diseases
* Any intracranial pathology present
* Surgeries exceeding 180 minutes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between the ages of 18-50 who will undergo total thyroidectomy under general anesthesia due to elective thyroid cancer, Hashimoto's thyroiditis or thyrotoxicosis, in the American Society of Anesthesiologists (ASA) I-II risk group, who are euthyroid in the preoperative period
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive functions | 3 months after surgery
  determine cognitive dysfunction using mini mental state examination

SECONDARY OUTCOMES:
Changes in Cerebral Perfusion | during surgery
  Changes in main carotid artery blood flow and cerebral oxygenation by using carotid doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No